CLINICAL TRIAL: NCT00117000
Title: The Effects of Testosterone and Nutritional Supplementation, Alone and Combined, on the Adverse Effects of Under-Nutrition in the Elderly
Brief Title: The Effects of Testosterone and Nutritional Supplementation in the Undernourished Elderly
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Adelaide (Other)
Collaborators: Organon (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 030320
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Malnutrition; Aging
Keywords: testosterone; food, formulated; malnutrition; undernutrition; aging; aged; aged, 80 and over; frail elderly
MeSH Terms: conditions — Malnutrition | interventions — testosterone undecanoate

INTERVENTIONS:
Drug: testosterone undecanoate

SUMMARY:
The purpose of this study is to determine what effect treatment for one year with testosterone and a nutritional supplement, alone and combined, has on the adverse effects of under-nutrition in community-dwelling older men and women.

DETAILED DESCRIPTION:
We hypothesize that oral androgen therapy and nutritional supplementation will have additive beneficial effects in older malnourished individuals living in the community; there will be a reduction in hospitalizations, falls and weight loss in association with improvements in functional measures and increases in lean body mass. The present study is designed to examine the effect of 12 months oral nutrition supplementation and androgen therapy, alone and combined, on (i) frequency and length of hospitalisations; (ii) functional status; (iii) body composition and weight; (iv) living arrangements; (v) death rate, in community dwelling under-nourished men and women, 65 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 years or older who are under-nourished, as defined by a Mini Nutritional Assessment (MNA) score <24 AND 1 or more of the following: *a body mass index (BMI) of less than 22 kg/m2; *weight loss of > 7.5% in the 3 months before enrolling in the study
* Living independently in the community (not in a hospital, nursing home or hostel)
* Understand and sign informed consent document, able to communicate with the investigator, and understand and comply with the requirements of the study.
* Women who are taking oestrogen or other hormone replacement therapy (HRT) may take part (see exclusion criteria for exceptions), as may women who are not taking HRT. If a woman is taking HRT she must have been on a stable dose for at least 3 months before enrolment in the study. If not on HRT, she must not have been taking it for at least 3 months before enrolment.

Exclusion Criteria:

* Dementia as indicated by a Folstein's Mini Mental State Examination (MMSE) score of < 23
* Elevated haematocrit (HCT) levels (>50%)
* Past or present history of prostatic cancer in men (Prostate Specific Antigen (PSA) levels [> age-related normal range and/or irregular prostate on prostate examination]) or breast cancer.
* Pre-existing androgenic signs or symptoms in women of concern to either subject or investigator (deep voice, hirsutism, acne, androgenic hair loss).
* Depression (Yesavage Geriatric Depression Scale (GDS) Score > 11)
* Inability to attend DEXA scan or complete other requirements of the study
* Significant cardiac failure (NYHA Class III and above)
* Significantly abnormal liver function tests (ALT, GGT, bilirubin or ALP more than 2 times the upper limit of normal)
* Nephrotic syndrome; 24h urine protein excretion > 3 grams (if baseline urinalysis reveals > 1+ proteinuria, quantification will be performed) AND/OR calculated creatinine clearance (by the equation of Baracskay and Jarjoura for ambulatory elderly subjects [Cr clearance = 4.4/serum creatinine (mmol/L) + (88-age)](63) < 30 ml/min) AND/OR serum creatinine concentration > 0.2mmol/l.
* Amputee (body mass index, creatinine clearance and body composition estimations inaccurate).
* Any disease, which in the opinion of the investigator is likely to lead to death within one year
* Testosterone or other androgen therapy (including DHEA and tibolone) in the four months before starting the study.
* Medication with cyclosporin or barbiturates

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200
Dates: Start 2003-07; Study Completion 2007-02

PRIMARY OUTCOMES:
Days in hospital
SF-36 quality of life scores (composite physical component score and composite mental component score).

SECONDARY OUTCOMES:
Body composition
Muscle strength
Number of falls
Functional status (living arrangements, activities of daily living and frailty scale scores)
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Chapman, MBBS, PhD, Principal Investigator — University of Adelaide
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Evans WJ, Campbell WW. Sarcopenia and age-related changes in body composition and functional capacity. J Nutr. 1993 Feb;123(2 Suppl):465-8. doi: 10.1093/jn/123.suppl_2.465. PMID 8429405
- [Background] Tenover JS. Androgen replacement therapy to reverse and/or prevent age-associated sarcopenia in men. Baillieres Clin Endocrinol Metab. 1998 Oct;12(3):419-25. doi: 10.1016/s0950-351x(98)80153-5. PMID 10332563
- [Background] Roshan S, Nader S, Orlander P. Review: Ageing and hormones. Eur J Clin Invest. 1999 Mar;29(3):210-3. doi: 10.1046/j.1365-2362.1999.00436.x. PMID 10202377
- [Background] Volpi E, Sheffield-Moore M, Rasmussen BB, Wolfe RR. Basal muscle amino acid kinetics and protein synthesis in healthy young and older men. JAMA. 2001 Sep 12;286(10):1206-12. doi: 10.1001/jama.286.10.1206. PMID 11559266
- [Background] Newman AB, Yanez D, Harris T, Duxbury A, Enright PL, Fried LP; Cardiovascular Study Research Group. Weight change in old age and its association with mortality. J Am Geriatr Soc. 2001 Oct;49(10):1309-18. doi: 10.1046/j.1532-5415.2001.49258.x. PMID 11890489
- [Background] MacIntosh C, Morley JE, Chapman IM. The anorexia of aging. Nutrition. 2000 Oct;16(10):983-95. doi: 10.1016/s0899-9007(00)00405-6. No abstract available. PMID 11054605
- [Background] Morley JE. Anorexia in older persons: epidemiology and optimal treatment. Drugs Aging. 1996 Feb;8(2):134-55. doi: 10.2165/00002512-199608020-00007. PMID 8845587
- [Background] Visvanathan R, Macintosh C, Callary M, Penhall R, Horowitz M, Chapman I. The nutritional status of 250 older Australian recipients of domiciliary care services and its association with outcomes at 12 months. J Am Geriatr Soc. 2003 Jul;51(7):1007-11. doi: 10.1046/j.1365-2389.2003.51317.x. PMID 12834523
- [Background] Morley JE. Testosterone replacement and the physiologic aspects of aging in men. Mayo Clin Proc. 2000 Jan;75 Suppl:S83-7. PMID 10959223
- [Background] Melton LJ 3rd, Khosla S, Riggs BL. Epidemiology of sarcopenia. Mayo Clin Proc. 2000 Jan;75 Suppl:S10-2; discussion S12-3. PMID 10959209
- [Background] Roubenoff R, Rall LC, Veldhuis JD, Kehayias JJ, Rosen C, Nicolson M, Lundgren N, Reichlin S. The relationship between growth hormone kinetics and sarcopenia in postmenopausal women: the role of fat mass and leptin. J Clin Endocrinol Metab. 1998 May;83(5):1502-6. doi: 10.1210/jcem.83.5.4809. PMID 9589646
- [Background] Davis S. Androgen replacement in women: a commentary. J Clin Endocrinol Metab. 1999 Jun;84(6):1886-91. doi: 10.1210/jcem.84.6.5802. PMID 10372681
- [Background] Zumoff B, Strain GW, Miller LK, Rosner W. Twenty-four-hour mean plasma testosterone concentration declines with age in normal premenopausal women. J Clin Endocrinol Metab. 1995 Apr;80(4):1429-30. doi: 10.1210/jcem.80.4.7714119.
- [Background] Burger HG, Dudley EC, Cui J, Dennerstein L, Hopper JL. A prospective longitudinal study of serum testosterone, dehydroepiandrosterone sulfate, and sex hormone-binding globulin levels through the menopause transition. J Clin Endocrinol Metab. 2000 Aug;85(8):2832-8. doi: 10.1210/jcem.85.8.6740. PMID 10946891
- [Background] Morley JE. Testosterone replacement in older men and women. J Gend Specif Med. 2001;4(2):49-53. PMID 11480098
- [Background] Morley JE. Androgens and aging. Maturitas. 2001 Feb 28;38(1):61-71; discussion 71-3. doi: 10.1016/s0378-5122(00)00192-4. PMID 11311591
- [Background] Davis SR, Burger HG. The rationale for physiological testosterone replacement in women. Baillieres Clin Endocrinol Metab. 1998 Oct;12(3):391-405. doi: 10.1016/s0950-351x(98)80115-8. PMID 10332561
- [Background] Tenover JL. Testosterone replacement therapy in older adult men. Int J Androl. 1999 Oct;22(5):300-6. doi: 10.1046/j.1365-2605.1999.00184.x. PMID 10509230
- [Background] Ly LP, Jimenez M, Zhuang TN, Celermajer DS, Conway AJ, Handelsman DJ. A double-blind, placebo-controlled, randomized clinical trial of transdermal dihydrotestosterone gel on muscular strength, mobility, and quality of life in older men with partial androgen deficiency. J Clin Endocrinol Metab. 2001 Sep;86(9):4078-88. doi: 10.1210/jcem.86.9.7821. PMID 11549629
- [Background] Amory JK, Chansky HA, Chansky KL, Camuso MR, Hoey CT, Anawalt BD, Matsumoto AM, Bremner WJ. Preoperative supraphysiological testosterone in older men undergoing knee replacement surgery. J Am Geriatr Soc. 2002 Oct;50(10):1698-701. doi: 10.1046/j.1532-5415.2002.50462.x. PMID 12366624
- [Background] Bakhshi V, Elliott M, Gentili A, Godschalk M, Mulligan T. Testosterone improves rehabilitation outcomes in ill older men. J Am Geriatr Soc. 2000 May;48(5):550-3. doi: 10.1111/j.1532-5415.2000.tb05002.x. PMID 10811549
- [Background] Chakravarti S, Collins WP, Forecast JD, Newton JR, Oram DH, Studd JW. Hormonal profiles after the menopause. Br Med J. 1976 Oct 2;2(6039):784-7. doi: 10.1136/bmj.2.6039.784. PMID 974609
- [Background] Zumoff B, Rosenfeld RS, Strain GW, Levin J, Fukushima DK. Sex differences in the twenty-four-hour mean plasma concentrations of dehydroisoandrosterone (DHA) and dehydroisoandrosterone sulfate (DHAS) and the DHA to DHAS ratio in normal adults. J Clin Endocrinol Metab. 1980 Aug;51(2):330-3. doi: 10.1210/jcem-51-2-330. PMID 6447161
- [Background] Davis SR, McCloud P, Strauss BJ, Burger H. Testosterone enhances estradiol's effects on postmenopausal bone density and sexuality. Maturitas. 1995 Apr;21(3):227-36. doi: 10.1016/0378-5122(94)00898-h. PMID 7616872
- [Background] Davis SR, Tran J. Testosterone influences libido and well being in women. Trends Endocrinol Metab. 2001 Jan-Feb;12(1):33-7. doi: 10.1016/s1043-2760(00)00333-7. PMID 11137039
- [Background] Castelo-Branco C, Vicente JJ, Figueras F, Sanjuan A, Martinez de Osaba MJ, Casals E, Pons F, Balasch J, Vanrell JA. Comparative effects of estrogens plus androgens and tibolone on bone, lipid pattern and sexuality in postmenopausal women. Maturitas. 2000 Feb 15;34(2):161-8. doi: 10.1016/s0378-5122(99)00096-1. PMID 10714911
- [Background] Gruber DM, Sator MO, Kirchengast S, Joura EA, Huber JC. Effect of percutaneous androgen replacement therapy on body composition and body weight in postmenopausal women. Maturitas. 1998 Jun 17;29(3):253-9. doi: 10.1016/s0378-5122(98)00031-0. PMID 9699197
- [Background] Padero MC, Bhasin S, Friedman TC. Androgen supplementation in older women: too much hype, not enough data. J Am Geriatr Soc. 2002 Jun;50(6):1131-40. doi: 10.1046/j.1532-5415.2002.50273.x. PMID 12110078
- [Background] Lobo RA. Androgens in postmenopausal women: production, possible role, and replacement options. Obstet Gynecol Surv. 2001 Jun;56(6):361-76. doi: 10.1097/00006254-200106000-00022. PMID 11466487
- [Background] Westaby D, Ogle SJ, Paradinas FJ, Randell JB, Murray-Lyon IM. Liver damage from long-term methyltestosterone. Lancet. 1977 Aug 6;2(8032):262-3. PMID 69876
- [Background] Raisz LG, Wiita B, Artis A, Bowen A, Schwartz S, Trahiotis M, Shoukri K, Smith J. Comparison of the effects of estrogen alone and estrogen plus androgen on biochemical markers of bone formation and resorption in postmenopausal women. J Clin Endocrinol Metab. 1996 Jan;81(1):37-43. doi: 10.1210/jcem.81.1.8550780.
- [Background] Davis SR, Burger HG. Clinical review 82: Androgens and the postmenopausal woman. J Clin Endocrinol Metab. 1996 Aug;81(8):2759-63. doi: 10.1210/jcem.81.8.8768824. No abstract available.
- [Background] Burger HG, Hailes J, Menelaus M, Nelson J, Hudson B, Balazs N. The management of persistent menopausal symptoms with oestradiol-testosterone implants: clinical, lipid and hormonal results. Maturitas. 1984 Dec;6(4):351-8. doi: 10.1016/0378-5122(84)90008-2. PMID 6442755
- [Background] Burger H, Hailes J, Nelson J, Menelaus M. Effect of combined implants of oestradiol and testosterone on libido in postmenopausal women. Br Med J (Clin Res Ed). 1987 Apr 11;294(6577):936-7. doi: 10.1136/bmj.294.6577.936. No abstract available. PMID 3107663
- [Background] Miller K, Corcoran C, Armstrong C, Caramelli K, Anderson E, Cotton D, Basgoz N, Hirschhorn L, Tuomala R, Schoenfeld D, Daugherty C, Mazer N, Grinspoon S. Transdermal testosterone administration in women with acquired immunodeficiency syndrome wasting: a pilot study. J Clin Endocrinol Metab. 1998 Aug;83(8):2717-25. doi: 10.1210/jcem.83.8.5051. PMID 9709937
- [Background] Mortola JF, Yen SS. The effects of oral dehydroepiandrosterone on endocrine-metabolic parameters in postmenopausal women. J Clin Endocrinol Metab. 1990 Sep;71(3):696-704. doi: 10.1210/jcem-71-3-696. PMID 2144295
- [Background] Casson PR, Santoro N, Elkind-Hirsch K, Carson SA, Hornsby PJ, Abraham G, Buster JE. Postmenopausal dehydroepiandrosterone administration increases free insulin-like growth factor-I and decreases high-density lipoprotein: a six-month trial. Fertil Steril. 1998 Jul;70(1):107-10. doi: 10.1016/s0015-0282(98)00121-6. PMID 9660430
- [Background] Phillips E, Bauman C. Safety surveillance of esterified estrogens-methyltestosterone (Estratest and Estratest HS) replacement therapy in the United States. Clin Ther. 1997 Sep-Oct;19(5):1070-84. doi: 10.1016/s0149-2918(97)80060-4. PMID 9385494
- [Background] Barnhart KT, Freeman E, Grisso JA, Rader DJ, Sammel M, Kapoor S, Nestler JE. The effect of dehydroepiandrosterone supplementation to symptomatic perimenopausal women on serum endocrine profiles, lipid parameters, and health-related quality of life. J Clin Endocrinol Metab. 1999 Nov;84(11):3896-902. doi: 10.1210/jcem.84.11.6153. PMID 10566625
- [Background] Diamond P, Cusan L, Gomez JL, Belanger A, Labrie F. Metabolic effects of 12-month percutaneous dehydroepiandrosterone replacement therapy in postmenopausal women. J Endocrinol. 1996 Sep;150 Suppl:S43-50. PMID 8943786
- [Background] Shifren JL, Braunstein GD, Simon JA, Casson PR, Buster JE, Redmond GP, Burki RE, Ginsburg ES, Rosen RC, Leiblum SR, Caramelli KE, Mazer NA. Transdermal testosterone treatment in women with impaired sexual function after oophorectomy. N Engl J Med. 2000 Sep 7;343(10):682-8. doi: 10.1056/NEJM200009073431002. PMID 10974131
- [Background] Dobs AS, Nguyen T, Pace C, Roberts CP. Differential effects of oral estrogen versus oral estrogen-androgen replacement therapy on body composition in postmenopausal women. J Clin Endocrinol Metab. 2002 Apr;87(4):1509-16. doi: 10.1210/jcem.87.4.8362. PMID 11932273
- [Background] Myers LS, Dixen J, Morrissette D, Carmichael M, Davidson JM. Effects of estrogen, androgen, and progestin on sexual psychophysiology and behavior in postmenopausal women. J Clin Endocrinol Metab. 1990 Apr;70(4):1124-31. doi: 10.1210/jcem-70-4-1124. PMID 1690746
- [Background] Watts NB, Notelovitz M, Timmons MC, Addison WA, Wiita B, Downey LJ. Comparison of oral estrogens and estrogens plus androgen on bone mineral density, menopausal symptoms, and lipid-lipoprotein profiles in surgical menopause. Obstet Gynecol. 1995 Apr;85(4):529-37. doi: 10.1016/0029-7844(94)00448-m. PMID 7898828
- [Background] Penotti M, Sironi L, Cannata L, Vigano P, Casini A, Gabrielli L, Vignali M. Effects of androgen supplementation of hormone replacement therapy on the vascular reactivity of cerebral arteries. Fertil Steril. 2001 Aug;76(2):235-40. doi: 10.1016/s0015-0282(01)01923-9. PMID 11476766
- [Background] Morley JE. Anorexia of aging: physiologic and pathologic. Am J Clin Nutr. 1997 Oct;66(4):760-73. doi: 10.1093/ajcn/66.4.760. PMID 9322549
- [Background] Mathey MF, Siebelink E, de Graaf C, Van Staveren WA. Flavor enhancement of food improves dietary intake and nutritional status of elderly nursing home residents. J Gerontol A Biol Sci Med Sci. 2001 Apr;56(4):M200-5. doi: 10.1093/gerona/56.4.m200. PMID 11283191
- [Background] Rolls BJ, McDermott TM. Effects of age on sensory-specific satiety. Am J Clin Nutr. 1991 Dec;54(6):988-96. doi: 10.1093/ajcn/54.6.988. PMID 1957832
- [Background] Ritchie CS, Burgio KL, Locher JL, Cornwell A, Thomas D, Hardin M, Redden D. Nutritional status of urban homebound older adults. Am J Clin Nutr. 1997 Oct;66(4):815-8. doi: 10.1093/ajcn/66.4.815. PMID 9322555
- [Background] Omran ML, Morley JE. Assessment of protein energy malnutrition in older persons, Part II: Laboratory evaluation. Nutrition. 2000 Feb;16(2):131-40. doi: 10.1016/s0899-9007(99)00251-8. PMID 10696638
- [Background] Lumbers M, New SA, Gibson S, Murphy MC. Nutritional status in elderly female hip fracture patients: comparison with an age-matched home living group attending day centres. Br J Nutr. 2001 Jun;85(6):733-40. doi: 10.1079/bjn2001350. PMID 11430778
- [Background] Middleton MH, Nazarenko G, Nivison-Smith I, Smerdely P. Prevalence of malnutrition and 12-month incidence of mortality in two Sydney teaching hospitals. Intern Med J. 2001 Nov;31(8):455-61. doi: 10.1046/j.1445-5994.2001.00109.x. PMID 11720058
- [Background] Sullivan DH, Walls RC, Lipschitz DA. Protein-energy undernutrition and the risk of mortality within 1 y of hospital discharge in a select population of geriatric rehabilitation patients. Am J Clin Nutr. 1991 Mar;53(3):599-605. doi: 10.1093/ajcn/53.3.599. PMID 1900382
- [Background] Abbasi AA, Rudman D. Undernutrition in the nursing home: prevalence, consequences, causes and prevention. Nutr Rev. 1994 Apr;52(4):113-22. doi: 10.1111/j.1753-4887.1994.tb01403.x. PMID 8028816
- [Background] de Jong N, Chin A Paw MJ, de Groot LC, de Graaf C, Kok FJ, van Staveren WA. Functional biochemical and nutrient indices in frail elderly people are partly affected by dietary supplements but not by exercise. J Nutr. 1999 Nov;129(11):2028-36. doi: 10.1093/jn/129.11.2028. PMID 10539780
- [Background] Lauque S, Arnaud-Battandier F, Mansourian R, Guigoz Y, Paintin M, Nourhashemi F, Vellas B. Protein-energy oral supplementation in malnourished nursing-home residents. A controlled trial. Age Ageing. 2000 Jan;29(1):51-6. doi: 10.1093/ageing/29.1.51. PMID 10690696
- [Background] Gray-Donald K, Payette H, Boutier V, Page S. Evaluation of the dietary intake of homebound elderly and the feasibility of dietary supplementation. J Am Coll Nutr. 1994 Jun;13(3):277-84. doi: 10.1080/07315724.1994.10718409. PMID 8077577
- [Background] Tkatch L, Rapin CH, Rizzoli R, Slosman D, Nydegger V, Vasey H, Bonjour JP. Benefits of oral protein supplementation in elderly patients with fracture of the proximal femur. J Am Coll Nutr. 1992 Oct;11(5):519-25. doi: 10.1080/07315724.1992.10718256. PMID 1452950
- [Background] Delmi M, Rapin CH, Bengoa JM, Delmas PD, Vasey H, Bonjour JP. Dietary supplementation in elderly patients with fractured neck of the femur. Lancet. 1990 Apr 28;335(8696):1013-6. doi: 10.1016/0140-6736(90)91073-j. PMID 1970070
- [Background] Schurch MA, Rizzoli R, Slosman D, Vadas L, Vergnaud P, Bonjour JP. Protein supplements increase serum insulin-like growth factor-I levels and attenuate proximal femur bone loss in patients with recent hip fracture. A randomized, double-blind, placebo-controlled trial. Ann Intern Med. 1998 May 15;128(10):801-9. doi: 10.7326/0003-4819-128-10-199805150-00002. PMID 9599191
- [Background] Sullivan DH, Patch GA, Walls RC, Lipschitz DA. Impact of nutrition status on morbidity and mortality in a select population of geriatric rehabilitation patients. Am J Clin Nutr. 1990 May;51(5):749-58. doi: 10.1093/ajcn/51.5.749. PMID 2110413
- [Background] Baracskay D, Jarjoura D, Cugino A, Blend D, Rutecki GW, Whittier FC. Geriatric renal function: estimating glomerular filtration in an ambulatory elderly population. Clin Nephrol. 1997 Apr;47(4):222-8. PMID 9128788
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Reuben DB, Siu AL. An objective measure of physical function of elderly outpatients. The Physical Performance Test. J Am Geriatr Soc. 1990 Oct;38(10):1105-12. doi: 10.1111/j.1532-5415.1990.tb01373.x. PMID 2229864
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Mazess RB, Barden HS, Bisek JP, Hanson J. Dual-energy x-ray absorptiometry for total-body and regional bone-mineral and soft-tissue composition. Am J Clin Nutr. 1990 Jun;51(6):1106-12. doi: 10.1093/ajcn/51.6.1106. PMID 2349926
- [Derived] Chapman IM, Visvanathan R, Hammond AJ, Morley JE, Field JB, Tai K, Belobrajdic DP, Chen RY, Horowitz M. Effect of testosterone and a nutritional supplement, alone and in combination, on hospital admissions in undernourished older men and women. Am J Clin Nutr. 2009 Mar;89(3):880-9. doi: 10.3945/ajcn.2008.26538. Epub 2009 Jan 14. PMID 19144729